CLINICAL TRIAL: NCT04143893
Title: SMart Angioplasty Research Team: A Multi-centeR, prospEctive Observational Study to Investigate the Current Status and Clinical oUtcomes of Patients With cardiogEnic Shock II: SMART-RESCUE II
Brief Title: The Current Status and Clinical Outcomes of Patients With Cardiogenic Shock II
Acronym: RESCUE II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Other Study IDs: RESCUEII
Record Dates: First submitted 2019-10-23; First posted 2019-10-29 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic shock; Mechanical Circulatory Support
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiogenic shock with MCS: Patients with cardiogenic shock who underwent MCS
  Interventions: Device: Mechanical circulatory support; Drug: Optimal medical treatment
- Cardiogenic shock without MCS: Patients with cardiogenic shock who did not undergo MCS
  Interventions: Drug: Optimal medical treatment

INTERVENTIONS:
Device: Mechanical circulatory support — Patients with cardiogenic shock who underwent MCS
  Groups: Cardiogenic shock with MCS
Drug: Optimal medical treatment — Patients with cardiogenic shock who received optimal medical treatment including vasopressor

SUMMARY:
The investigation of patient characteristics and prognostic factors of the patients presented with cardiogenic shock (CS) will guide us to identify the better management strategy for these critically ill patients. Mechanical circulatory support (MCS) may improve the prognosis of some of severe subset of CS patients. The better understanding of the indications of initiation and weaning of MCS will improve the prognosis of critically ill CS patients.

DETAILED DESCRIPTION:
Patients presented with cardiogenic shock (CS) still have a very poor prognosis with high in-hospital mortality even in current era of medical practice. Acute myocardial infarction (AMI) complicated by CS has been associated with is an in-hospital survival of around 50% historically. Recent development of mechanical circulatory support (MCS) showed a better survival in the patients who would have been associated with a very high mortality in conventional medical treatment. Still the most of the management strategy for this critically ill patient subset is empirical and mostly not based on scientific evidence. There have been few randomized controlled trials and well-designed registries have been rare.

Recent randomized controlled trial, IABP SHOCK II trial showed that use of IABP did not improve survival in CS patients complicating AMI. With the FDA approval of Impella in CS patients, a powerful new tool has become available for hemodynamic support. Impella is a transcatheter axial flow pump, delivered percutaneous, with the ability to provide 2.5 to 4.0 liters/minute of forward flow. In some countries where Impella is not available, extracorporeal membrane oxygenator (ECMO) has been widely used in patients with cardiac arrest or CS. ECMO is equipped with an oxygenator and may be more beneficial in the patients with cardiac and pulmonary failure. Impella is a more physiological device that does not compete with native blood flow. However, there is little data available to providers as to the best practice patterns associated with the delivery and use of mechanical circulatory devices in CS patients, furthermore, no data regarding CS patients originated by non-ischemic and post-cardiotomy situation as an etiology of cardiogenic shock.

Around 20 years ago, it is conducted CS registry and then, Cardshock registry launched in 2010 and enrolled only 219 patients. Well-designed large scale registries of CS patients are scarce. Recently, the investigators conducted retrospective and prospective registry of patient with cardiogenic shock (RESCUE I registry) and just finished to enroll 1247 patients from 12 centers in Korea between January 2014 and December 2018. ECMO device was used in 496 patients (40%) and IABP was used in 298 patients (24%). The registry is under analysis to investigate clinical characteristics and predictors of in-hospital mortality. The major weakness of RESCUE I registry are ;1) major proportion of the patients were enroll retrospectively, 2) the etiology of shock was not well defined, and most of enrolled population were of ischemic etiology, 3) the variables in the case record form was not systematically structured. Based on the RESCUE I registry, the investigators would like to launch RESCUE II registry as an prospective registry with well-defined subgroups of ischemic, myocardial, post-cardiotomy etiologies, and more systematically arranged variables based on prospective protocols or guidelines of management based on RESCUE I registry.

The investigators believe that the differences of races, management, and difference types of MCS can influence the outcomes of CS patients, but still there were no evidence. Mayo clinic is one of the top medical centers of excellence with experiences and science in the field of critically ill patients. The collaboration of Mayo Clinic team and RESCUE research team in Korea will be quite synergistic by sharing their knowledge and experience in the management and research in this filed.

The ultimate goal of RESCUE II is to develop the evidence-based medicine for the patients with cardiogenic shock by bringing experienced centers together across the 2 nations who are experts in mechanical circulatory support devices as well as the medical management in critically ill CS patients. The investigators aim to find optimal monitoring strategy, medical management, as well as best protocols for the application of mechanical circulatory support.

ELIGIBILITY:
Inclusion Criteria:

* 19 years old or older
* Cardiogenic shock is defined as the presence of the following:

  1. Systolic blood pressure is less than 90mmHg for more than 30 minutes despite the fluid therapy, or the use of pressure boosting agents to maintain the systolic blood pressure more than 90 mmHg.
  2. Peripheral hypoperfusion (cold skin, urine less than 30 cc per hour, impaired consciousness, lactate ≥2.0 mmol/l) or a person with pulmonary edema.
* Causes of cardiogenic shock include ischemic (acute myocardial infarction or ischemic cardiomyopathy, shock during cardiac intervention), myocardial (end-stage heart failure, myocarditis), post-cardiotomy shock, cardiac tamponade, or pulmonary thromboembolism.
* Those voluntarily consenting to the medical records and the data necessary for the study during the entire study period.

Exclusion Criteria:

* Other causes except for cardiogenic shock: septic shock, cardiac arrest by serious ventricular arrhythmia not related to the myocardial ischemia or heart failure
* Shock with unwitnessed cardiac arrest outside the hospital
* Severe non-cardiac morbidity with expected survival less than 6 months (malignancy, respiratory failure)
* Those who refused active treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 1000 patient with cardiogenic shock
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital all-cause mortality | Up to 12 weeks
  Death in-hospital

SECONDARY OUTCOMES:
In-hospital cardiac mortality | Up to 12 weeks
  Cardiac death in-hospital
In-hospital neurologic outcome | Up to 12 weeks
  Defined by the cerebral performance category (CPC) scoring system (ranges from 1 to 5 / good outcome as a CPC score of 1 or 2, and a poor outcome [severe neurological disability, persistent vegetative state or death] as CPC scores 3, 4, or 5)
Death in 30days | 30 Days after admission
  30 Days mortality
Cardiac death in 30 days | 30 Days after admission
  30 Days cardiac mortality
MACE | through study completion, an average of 1 year
  Death, myocardial infarction, stroke, re-admission due to heart failure, and heart transplantation during follow-up.
Lactate clearance | 24 hours after admission
  Lactate 24 hour clearance
Successful weaning of mechanical circulatory support device | Up to 12 weeks
  In-hospital successful weaning of mechanical circulatory support device, including IABP, Impella, and ECMO. (successful weaning or failed weaning)

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea